CLINICAL TRIAL: NCT03997591
Title: Effect of Ready2E.A.T. in Risk Populations
Brief Title: Upper Limb Reeducation Across Life Span
Acronym: ULReed
Status: Completed | Type: Observational
Sponsor: Instituto Politécnico de Leiria (Other)
Responsible Party: Principal Investigator, Marlene Rosa, Clinical Professor, Instituto Politécnico de Leiria
Other Study IDs: IPL10062019
Record Dates: First submitted 2019-06-10; First posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Upper Extremity Dysfunction; Dementia; Cerebral Palsy; Cognitive Decline; Eating Disorders
Keywords: eating; upper limb; reeducation
MeSH Terms: conditions — Dementia; Cerebral Palsy; Cognitive Dysfunction; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional therapy: Group doing conventional rehabilitation was assessed at T0 and then after 6 weeks of conventional therapy (occupational therapy, physical therapy, aquatic therapy, musicotherapy, others)
  Interventions: Other: Ready2E.A.T. PROGRAM
- Ready2E.A.T. therapy: Group doing Ready2E.A.T. program received a mean of 1 hour per week and was assessed at T0 and then after 6 weeks of this program implementation.
  Interventions: Other: Ready2E.A.T. PROGRAM

INTERVENTIONS:
Other: Ready2E.A.T. PROGRAM — Training tasks based on:
  reaching activities during attention tasks, memory tasks, sequential tasks This group was assessed at T0 and then after 6 weeks of conventional therapy.

SUMMARY:
Program Ready2E.A.T. was developed to be tested in the upper limb reeducation on population at risk, such as:

* Children with dysfunction
* Cognitive impaired elderly
* Dementia people

DETAILED DESCRIPTION:
Program Ready2E.A.T. consists on the training of specific upper limb tasks, including:

* reaching during attention tasks
* reaching during memory tasks
* reaching during sequential motor tasks
* reaching during fine hand movements

This program has been tested as a measure of functional status (cognitive and motor habilities) in population with different risks; It also has been tested as an effective program for reeducation in cognitive affected population.

ELIGIBILITY:
Inclusion Criteria:

* people with 60years old with cognitive decline
* children aging 6-10 years old with cognitive and motor dysfunction
* dysfunction in feeding participation

Exclusion Criteria:

* participants that do not understand 2 simnultaneous verbal commands

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Old people and children dependent in feeding activity.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

PRIMARY OUTCOMES:
Video analysis of feeding performance | 6 weeks
  performance of several feeding steps

SECONDARY OUTCOMES:
Frontal assessment battery | 6 weeks
  Assessment of Executive Functions

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Politécnico de Leiria, Leiria, Portugal

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT03997591/SAP_000.pdf